CLINICAL TRIAL: NCT00279734
Title: An Exploratory Study to Evaluate the Effect of Abatacept (BMS-188667) on the Antibody Response Following Tetanus Toxoid and 23-Valent Pneumococcal Vaccinations in Healthy Subjects
Brief Title: Vaccination Study of Abatacept (BMS-188667) for Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM101-049
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tetanus Toxoid; Abatacept; Vaccines

ARMS (4):
- Group 1 (Experimental)
  Interventions: Drug: Tetanus + pnemococcal vaccines alone
- Group 2 (Active Comparator)
  Interventions: Drug: Abatacept + vaccines
- Group 3 (Active Comparator)
  Interventions: Drug: Abatacept + vaccines
- Group 4 (Active Comparator)
  Interventions: Drug: Abatacept + Vaccines

INTERVENTIONS:
Drug: Tetanus + pnemococcal vaccines alone — 0 mg + vaccines, Single dose, 28 days.
  Arms: Group 1
Drug: Abatacept + vaccines — Parenteral, IV, 750 mg abatacept + vaccines, Single dose, 70 days.
  Other Names: Orencia
  Arms: Group 2
Drug: Abatacept + vaccines — Parenteral, IV, 750 mg abatacept + vaccines, Single dose, 56 days.
  Other Names: Orencia
  Arms: Group 3
Drug: Abatacept + Vaccines — parenteral, IV, 750 mg abatacept + vaccines, Single dose, 84 days.
  Other Names: Orencia
  Arms: Group 4

SUMMARY:
Study to assess the ability of healthy subjects to build anitbodies to tetanus and pneumococcal vaccines after receiving a single intravenous dose of Abatacept, a drug which is being developed for the treatment of Rheumatoid Arthritis and which can affect the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects
* Body Weight between 60 and 100 kg.
* Males and Females must be using adequate contraceptive methods during study and for 10 weeks after dose of study mediciation.

Exclusion Criteria:

* Females who are prgnant or breastfeeding
* History of autoimmune disorder, immunodeficiency, or infection within past 3 months.
* Active TB requiring treatment within the previous 3 years.
* Positive breast cancer screen, PPD test.
* Vaccination with tetanus or pneumococcal vaccine within 5 years.
* Vaccination with any live vaccine within 4 weeks.
* History of drug or alcohol abuse.
* Any significant allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-08; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Assess effect of single 750mg dose of Abatacept on antibody response to tetanus toxioid and 23-valent pneumococcal vaccines.

SECONDARY OUTCOMES:
Assess safety and tolerability of Abatacept given in conjunction with tetanus toxoid and 23-valent pneumococcal vaccines.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Qutintiles Phase I Services, Lenexa, Kansas
  - Parexel International Corp, Baltimore, Maryland
  - PPD Development, Austin, Texas

REFERENCES:
- [Derived] Tay L, Leon F, Vratsanos G, Raymond R, Corbo M. Vaccination response to tetanus toxoid and 23-valent pneumococcal vaccines following administration of a single dose of abatacept: a randomized, open-label, parallel group study in healthy subjects. Arthritis Res Ther. 2007;9(2):R38. doi: 10.1186/ar2174. PMID 17425783